CLINICAL TRIAL: NCT00125086
Title: Platelets in Acute Wounds: A Punch Biopsy Study (PAWS II)
Brief Title: Platelets for Acute Wound Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: APG-01-0605; APG-01-0605
Record Dates: First submitted 2005-07-27; First posted 2005-07-29 (Estimated); Last update posted 2005-09-14 (Estimated); Status verified 2005-09

CONDITIONS: Wounds
Keywords: wounds; healing; Acute wounds healing by secondary intention
MeSH Terms: conditions — Wounds and Injuries

INTERVENTIONS:
Device: autologous platelet gel

SUMMARY:
This study will examine whether platelet gel positively affects wound healing. Platelet gel will be used to treat punch biopsy wounds and the results will be compared to results from wounds treated with a control treatment.

DETAILED DESCRIPTION:
Platelets contribute to the healing process in soft tissue by providing the initial hemostasis that occurs following injury, a framework for fibrin matrix formation and contribution of growth factors.

According to the US National Institutes of Health, surgical procedures are considered a form of controlled injury, so many of the complications faced by surgery patients are very similar to those faced by trauma patients. Scientists are currently investigating ways to treat wounds caused by trauma, burns or surgical inventions with biological agents (i.e. growth factors) or new drugs. Growth factor priming of acute wound sites pre-activates the cellular and molecular components of tissue repair, prior to tissue injury.

Objectives are aimed at gathering information to establish evidence that autologous platelet gel positively effects the healing of acute wounds.

ELIGIBILITY:
Inclusion Criteria:

* Normal volunteers
* 18 years old or older

Exclusion Criteria:

* Pregnant or lactating
* Diabetic, keloid former, collagen vascular disease
* Smoker
* Body mass index >30kg/m2
* Known history of HIV/AIDS; Hepatitis A, B, or C
* Bleeding disorder
* Aspirin, non-steroidal anti-inflammatory drug (NSAID) or anticoagulant user
* Cancer, or treatment for cancer, in past 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4
Dates: Start 2005-07; Study Completion 2006-02

PRIMARY OUTCOMES:
Time to 100% wound closure, measured at Days 7, 14, 21, 28, 35

SECONDARY OUTCOMES:
Measurements of wound depth at each visit
Measurement of residual scarring at 6 months post wounding

CONTACTS AND LOCATIONS:
Overall Officials: David Hom, M.D., Principal Investigator — University of Minnesota
Locations (1):
- DaVita Clinical Research, Minneapolis, Minnesota, United States